CLINICAL TRIAL: NCT05946915
Title: The Use of miRNA Panel as a Growth Plate Marker of Short-term Response to GH
Brief Title: miRNA as a Growth Plate Marker After GH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Faculdade de Ciências Médicas da Santa Casa de São Paulo (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Carlos Alberto Longui, Full Professor, Faculdade de Ciências Médicas da Santa Casa de São Paulo
Other Study IDs: 67005222.0.0000.5479
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: MicroRNAs: D13.444.735.790.552.500

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The therapeutic use of recombinant human growth hormone usually determines adequate growth response in the majority of approved conditions. However, it is well recognized an inter-individual responsiveness, and the classical biomarker such as GH peak response, IGF-I or IGFBP3 levels have poor correlation with clinical outcome. We hypothesize that markers directed originated from the growth plate would have the potential to better correlate with growth response during GH treatment. Genetic markers, as the growth hormone receptor exon 3-deletion polymorphism, IGFBP3 polymorphisms were previously tested in an attempt to discriminate the pattern of responsiveness, but results were contradictory in the different studies. MicroRNAs (miRNAs) are small non-coding RNAs that regulate gene expression. Due to their ability to regulate gene expression, miRNAs play an important role both in physiology and pathophysiological conditions, and also an important role in the regulation of endochondral ossification and regulation of the hypothalamic-pituitary-IGF axis. Several miRNAs are already recognized as involved in the regulation of longitudinal growth and bone development, through its action upon WNT-βcatenin, Notch, PI3K/AKT and TGFβ signaling pathways. AIM: Therefore, the aim of this study is to establish a panel of miRNAs correlated to the growth response during GH treatment, that can be used of biomarker for early recognition and classification of patients according to GH therapy responsiveness. This study will analyze 30 Children and adolescents with GH deficiency associated with Ectopic Posterior Pituitary (EPP) gland. METHODS: Clinical, biochemical and miRNAs concentration will be measured at four time-points: before starting therapy (basal), and after 1-, 3- and 6-months during GH treatment. Studied variables include: height, target height, growth velocity and body mass index, bone age and pubertal stage. Laboratory Assessment: at basal condition: fasting glucose, insulin, TSH and free T4; and cortisol, and IGF-I at 3 and 6 months. Bone age at basal and 6 months of therapy. MiRNAs will be measured in peripheral blood sample obtained before starting GH therapy, after 1-, 3- and 6-months during GH treatment. A miRNA panel will be measured by absolute quantitative method (digital PCR). The identification of a panel of miRNAs that correlates with GH responsiveness offers a huge clinical applicability, allowing prompt identification of patients who need differential therapeutic protocols targeted to achieve the best response during GH treatment.

DETAILED DESCRIPTION:
Introduction The clinical experience with the therapeutic use of recombinant human growth hormone (GH) has found adequate growth response in the majority of patients treated for each of the approved indications. However, as the experience accumulates with different treatment regimens, it was recognized that individual first-year height responses vary considerably even with individualized treatment regimens (1). Poor short-term response is also translated into an unsatisfactory gain in adult height (2).

Some mathematical models were developed in order to predict growth response of an individual patients. Prediction models derived from the large Pfizer International Growth Database (KIGS) database explain approximately 60% of the variability of response to GH therapy in patients with GHD (3). Such models account for the definable variability of responsiveness, allowing clinicians to adjust GH dose to individual patient. Based on multiple regression analyses, these models have identified factors that correlate with growth (mainly first year growth velocity), such as chronological age, GH peak during provocative tests, GH dose, birth-weight SDS, height SDS adjusted for target height SDS (3). Biochemical variables such as the baseline IGF-I and leptin have also been added to the prediction models.

Genetic markers were also used in an attempt to discriminate good and bad responders to GH treatment, as the exon 3-deleted growth hormone receptor polymorphism, IGFBP3 polymorphism and others, but their results were contradictory in the different studies.

MicroRNAs (miRNAs) are small non-coding RNAs that regulate gene expression. Most genes in the human genome are regulated by one or more miRNAs (4). Due to their ability to regulate gene expression, miRNAs appear to play an important role in the pathophysiology and development of physiological processes, as well as in human diseases (5). MicroRNAs usually suppress gene expression by binding to the 3'UTR domain of mRNA (6), therefore increasing mRNA degradation or preventing translational information and protein synthesis.

One of the remarkable characteristics of miRNAs is the plasma circulation inside exosomes, determining its resistance to degradation, allowing its measurement in the circulating blood, performing as a liquid biopsy (7).

Scientific evidence in different in-vitro models and in animals, suggested that miRNAs have an important role in the regulation of endochondral ossification and in the regulation of the hypothalamic-pituitary-IGF axis (8). In particular, miRNA-140, 322 and 22 have been described as responsible for growth plate development (9). Catellani et al, showed that miR-22-3p, miR-30c-5p, miR-106a-5p, miR-140-5p, miR-199a-5p, miR-335-5p, miR-340- 5p, and miR-494-3p are involved in the regulation of longitudinal growth and bone development, through its action upon WNT-βcatenin, Notch, PI3K/AKT and TGFβ signaling pathways (10).

Growth response in patients during GH treatment is variable, depending both on the patient's basal conditions and on individual innate sensitivity to therapy (11). Often, the measured growth rate does not coincide with the expected one and the degree of correlation between clinical-auxological parameters and dose and GH peak vary enormously, both inter and intra-individually during treatment (12).

Therefore, the aim of this study is to measure the circulating growth plate synthesized miRNAs before and during GH treatment, searching for its correlation with clinical and biochemical markers.

Methods Children and adolescents (n:30 patients), both genders, with GH deficiency (GHD) followed at the Pediatric Endocrinology Unit of the Irmandade da Santa Casa de Misericórdia de São Paulo, Brazil, will be screened. Written informed consent will be obtained from all participants and their parents as appropriate.

Inclusion Criteria: GH stimulation test showing GH-peak concentration <5ng/ml, combined to magnetic resonance imaging showing Posterior Pituitary Ectopic gland (EPP). Patients with combined hormone deficiencies must be compensated during the study period.

Exclusion criteria: chronic diseases, need of prolonged supraphysiologic doses of glucocorticoids, bone age >14 years or >16 years (girls and boys, respectively), patients missing adequate follow-up during the study protocol.

Clinical follow-up: Clinical records at each visit will include age, weight, height, height to target height difference and pubertal stage. Clinical evaluation will be taken at five time-points: before starting therapy (basal), and after 1-, 3- and 6-months during GH treatment. The body mass index (BMI) will be calculated as weight/height² (kg/m²). Height, target height (TH) and BMI will be expressed as a SD score (WHO, 2007). Growth velocity SDS will be calculated using Tanner reference (13). Puberty in all subjects will be classified following Marshall and Tanner's criteria (14, 15). The bone age was will be obtained every 6 months and classified according to Greulich and Pyle (16).

Laboratory Assessment: Hormone measurements will be measured at 3 and 6 months and will include IGF-I, fasting glucose, insulin, TSH and free T4; and cortisol. Gonadotropins and sex steroids will be measured when adequate. To evaluate the expression of growth plate synthesized miRNAs, a basal blood sample will be obtained before starting GH therapy or after a short-time washout period (15-30 days) and after 1-, 3- and 6-months during GH treatment.

MiRNAs determination: quantitative PCR (qPCR) will be used to measure circulating miRNA levels, by employing the droplet digital PCR (ddPCR), considered to be the gold standard in the application of liquid biopsy, because its superior precision and sensitivity, being less affected by PCR inhibitors, and do not require internal/external normalization while detecting low concentration of target nucleic acids molecules. A whole blood sample will be drawn in vacutainer serum separator tubes, and processed within 2h from collection, centrifuged at 2,000 g for 10 min at 4°C. Serum will be aliquoted in 1.5-ml sterile RNase-free tubes and further centrifuged at 2,500 g for 10 min at 4°C to remove any contaminant cells and debris. Serum will be collected in sterile RNase-free tubes and stored at -80°C until use. Total RNA will be isolated from the sample using 200 ul of serum using the miRNeasy Serum/Plasma Advanced Kit (ID: 217204 - Qiagen).

The following miRNAs will be measured: miR-22-3p, miR-30c-5p, miR-106a-5p, miR-140-5p, miR-199a-5p, miR-335-5p, miR-340-5p, and miR-494-3p. For each ddPCR assay, 3 μL cDNA sample, 10 μL 2× ddPCR supermix for probes (Bio-Rad), 1 μL 20× TaqMan miRNA probe and 6 μL RNase-free Water will be added in a 20 μL reaction mixture. Then, the mixture and 70 μL droplet generation oil for probes (Bio-Rad) will be respectively loaded into the sample wells and oil wells of a disposable droplet generator cartridge (Bio-Rad). After that, droplets will be generated by QX200 droplet generator device (Bio-Rad) and carefully transferred to a 96-well PCR plate (Eppendorf). The cycling conditions will be: 95 °C for 10 min, 40 cycles of 95 °C for 15 s and 57 °C for 1 min, and a final step at 98 °C for 10 min. At the end of the PCR reaction, droplets will be read in the QX200 droplet reader and analyzed using the Quantasoft™ version 1.7.4 software (Bio-Rad).

Benefits: Establishing a panel of miRNAs that correlates with GH responsiveness is of huge clinical applicability, allowing prompt identification of patients who need differential therapeutic protocols targeted to achieve the best response during GH treatment.

ELIGIBILITY:
Inclusion Criteria:

* GH stimulation test showing GH-peak concentration <5ng/ml, combined to magnetic resonance imaging showing Posterior Pituitary Ectopic gland (EPP). Patients with combined hormone deficiencies must be compensated during the study period.

Exclusion Criteria:

* chronic diseases, need of prolonged supraphysiologic doses of glucocorticoids, bone age >14 years or >16 years (girls and boys, respectively), patients missing adequate follow-up

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Thirty patients with pituitary insufficiency related to Ectopic Posterior Pituitary gland
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-03 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Variation in microRNAs concentration | basal to six-months
  serial serum microRNAs concentration
Variation in height SDS | basal to six-months
  serial height SDS measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Santa Casa SP School of Medical Sciences, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pellicciari CR, Bispo TR, Rodart IF, Steinmetz L, Miachon AAS, Spinola E Castro AM, Damiani D, Kochi C, Longui CA. The Use of miRNA Panel as a Growth Plate Marker of Short-Term Response to GH. Clin Endocrinol (Oxf). 2025 Sep;103(3):327-337. doi: 10.1111/cen.15278. Epub 2025 May 20. PMID 40394920